CLINICAL TRIAL: NCT03623542
Title: Risk Factors for Adverse Drug Reactions in Older Subjects Hospitalized in a Dedicated Dementia Unit
Brief Title: Adverse Drug Reactions in Older Subjects
Acronym: RiskofADR
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2017Ao002
Record Dates: First submitted 2018-07-19; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Dementia
Keywords: Dementia; alzheimer dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dementia or alzheimer dementia: All patients presenting with dementia syndrome and whose admission was unplanned between May 2010 and November 2011 were consecutively included in the study.

SUMMARY:
Objective: To identify risk factors for the occurrence of adverse drug reactions (ADRs) based on geriatric evaluation.

Design: Longitudinal prospective study from May 2010 to November 2011. Setting: Dedicated acute geriatric care unit specializing in the management of patients with dementia at the University Hospital of Reims, France.

Measurements: Sociodemographic variables and comprehensive geriatric assessment were recorded. Occurrence of ADRs was noted. Risk factors for ADR were identified by multivariate logistic regression.

DETAILED DESCRIPTION:
Introduction: Adverse drug reactions (ADRs) are frequent among older subjects, and are actually avoidable in up to 60% of cases. There are few studies identifying the risk factors for ADRs based on comprehensive geriatric assessment in older subjects with dementia, although better identification of patients at risk could help to target patients at risk for increased morbidity and mortality due to ADRs with a view to taking appropriate preventive measures.

Objective: To identify risk factors for the occurrence of adverse drug reactions (ADRs) based on geriatric evaluation.

Design: Longitudinal prospective study from May 2010 to November 2011. Setting: Dedicated acute geriatric care unit specializing in the management of patients with dementia syndrome (Alzheimer disease or related syndromes) at the University Hospital of Reims, France.

Participants: Older patients with dementia syndrome (Alzheimer disease or related syndromes).

Measurements: Sociodemographic variables and comprehensive geriatric assessment were recorded. Occurrence of ADRs was noted. Risk factors for ADR were identified by multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia syndrome
* unplanned hospitalisation between may 2010 and november 2011

Exclusion Criteria:

- no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with dementia syndrome and whose admission was unplanned between May 2010 and November 2011 were consecutively included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-11-01 (Actual)

PRIMARY OUTCOMES:
Risk factors for the occurrence of adverse drug reactions | Month 18
  Factors (as comprehensive geriatric assessment : instrumental activities of daily living scale, Katz's activities of daily living scale, mini nutritional assessment short-form, mini mental state examination) associated with adverse drug reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Kanagaratnam L, Drame M, Novella JL, Trenque T, Joachim C, Nazeyrollas P, Jolly D, Mahmoudi R. Risk Factors for Adverse Drug Reactions in Older Subjects Hospitalized in a Dedicated Dementia Unit. Am J Geriatr Psychiatry. 2017 Mar;25(3):290-296. doi: 10.1016/j.jagp.2016.07.002. Epub 2016 Sep 1. PMID 27742527